CLINICAL TRIAL: NCT00727363
Title: Prophylactic Probiotics for the Prevention of Sepsis and NEC in Premature Infants in Colombia. A Randomized Double-Blind, Multicenter Trial
Brief Title: Prophylactic Probiotics in Premature Infants
Acronym: C3P
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: We are underpowered to find a difference in the primary outcome.
Sponsor: Colombian Neonatal Research Network (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); Vanderbilt University (Other)
Responsible Party: Mario Augusto Rojas MD, MPH, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CNRNProbiotics
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Death; Nosocomial Infection
Keywords: probiotics; lactobacillus reuteri; preterm infants; nosocomial infection; necrotizing enterocolitis
MeSH Terms: conditions — Death; Cross Infection; Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): 5 drops of an available oil suspension without Lactobacillus reuteri will be given once per day until discharge from the hospital. Patients fed through NG tube will be administered 5 drops of placebo through the NG tube followed by a 0.5 cc of a normal saline flush. Patients taking PO feeds will be administered 5 drops of placebo in posterior oropharynx after secretions have been suctioned.
  Interventions: Dietary Supplement: Placebo
- 2 (Experimental): 5 drops of Lactobacillus reuteri DSM 17938 from an oil based suspension will be administered once a day until death or discharge home. Patients with NG feeds will be administered the probiotic in the amount of 5 drops through the NG tube followed by 0.5 cc of a normal saline flush. Patients with PO feeds will be administered 5 drops of the probiotics in the posterior oropharynx after secretions have been suctioned. If feeds are temporarily suspended because of feeding intolerance or NEC, the probiotic may be re-started once feeds are re-started.
  Interventions: Dietary Supplement: Lactobacillus reuteri

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — Lactobacillus reuteri DSM 17938 will be administered at a dose of ten to the eighth colony-forming units in 5 drops of a commercially available oil suspension once per day until discharge from the hospital.
  Other Names: BioGaia Probiotic drops
  Arms: 2
Dietary Supplement: Placebo — 5 drops of an available oil suspension without Lactobacillus reuteri will be given once per day until discharge from the hospital.
  Arms: 1

SUMMARY:
This study tries to determine whether the oral administration of a specific probiotic (good bacteria) in premature infants hospitalized in a neonatal intensive care unit may prevent infections and the development of a severe inflammatory disease of the bowel called necrotizing enterocolitis. The investigators propose that premature infants not given probiotics will colonize their gut with bad bacterias and develop infection.

DETAILED DESCRIPTION:
Neonatal infections currently cause about 1.6 million deaths annually in developing countries. Preterm infants are especially vulnerable to infections because of their immature immune responses and their exposure to the hospital milieu which promotes gastrointestinal colonization with Gram-negative pathogens. Multiple studies have shown that the colonization of the bowel with probiotics (nonpathogenic anaerobic bacteria) competitively inhibit the attachment of Gram-negative pathogens decreasing their likelihood for bacterial translocation and the development of life threatening infections.This potentially high-impact, low-cost intervention may significantly improve the survival and morbidity of preterm infants around the world.

RESEARCH OBJECTIVE

We seek to determine whether prophylactic administration of Lactobacillus reuteri decreases the incidence of death and nosocomial sepsis among susceptible preterm infants in a neonatal care setting in Colombia.

Specific aims:

1. To investigate the efficacy and safety of oral Lactobacillus reuteri for the primary endpoint prevention of death or nosocomial sepsis in preterm infants through a well powered multicenter, randomized, double-blinded, placebo-controlled clinical trial (RCT).
2. To assess the impact of Lactobacillus reuteri on four secondary endpoints: necrotizing enterocolitis, prevalence of Gram-negative pathogens, duration of hospitalization, and frequency of outpatient treatment and re-admission for infectious causes at 6 months post-discharge.

RESEARCH DESIGN AND METHODS

Study Design:

Overview

Multi-center, double-blind, randomized, placebo-controlled trial Primary outcome: Death or nosocomial sepsis Secondary outcomes: NEC, prevalence of Gram-negative pathogens, duration of hospitalization, and frequency of outpatient treatment and re-admission for infectious causes at 6 months post-discharge. Post-hoc analysis will evaluate differences in RCT outcomes in two key subgroups: breast-fed and formula-fed infants and vaginal delivery versus cesarean section, in both probiotic exposed and unexposed infants. In addition, we will look at death and nosocomial sepsis as separate outcomes to ensure there is no differential effect of treatment in either outcome. Location: 11 NICUs in Colombia.

Randomization and Stratification:

Stratification according to participating institutions will be done in order to control for center-related differences. Stratification by birth weight will be performed in 2 groups: < 1500 grams and 1501 to 2000 grams. When eligibility criteria are met, infants will be randomly assigned to treatment with probiotics or placebo by using a computerized stratified balanced block randomization design. Assignment to treatment will be accomplished using sealed, sequentially numbered, opaque envelopes, color-coded for strata, available in each NICU pharmacy.

Experimental Design:

Study patients will be randomized at birth to either placebo or probiotic administration (treatment group). The hospital pharmacy will be in charge of random allocation. Vials of probiotic and placebo will only be identified by the pharmacist and according to randomization will be sent to the NICU for administration to the patient. For those randomized to the treatment arm, L reuteri DSM 17938 will be administered at a dose of 10 to the eighth colony-forming units in 5 drops of a commercially available oil suspension once per day until discharge from the hospital. This oil suspension is stable for 21 months at 2o C to 8o C (as documented by the manufacturer, BioGaia AB, Stockholm, Sweden). For those randomized to the placebo arm, patients will receive an equal number of drops from an identical vial containing only the oil base, but without the probiotic. The above preparations will be administered even if the patient has not begun a feeding protocol if there are no contraindications for feeding. Patients will be stratified according to their exposure to breast milk or premature infant formula alone or a combination of both. Infants of mothers with insufficient production of breast milk will be offered premature formula.

Feeding and nutrition protocols will be standardized among participating institutions to minimize the confounding effects of diverse practices. A standard feeding protocol may be started at 24-48 hours of life at a volume of 10 ml/kg/day if the patient is hemodynamically stable, defined as having a stable blood pressure. The two milliliters of breast milk or premature infant formula will be subtracted from this total daily volume. Feedings will be advanced slowly at a volume between 10 and 20 ml/kg/day depending on tolerance.84 Umbilical lines may be removed once feeds are increased above 20 ml/kg/day. Parenteral nutrition will be started on the second day of life according to a standardized protocol. MCT oil (2 kcal/30ml) will be used as a dietary supplement to increases the energy content of breast milk or formula when needed. Human milk fortifiers may be started once full enteral feeds have been tolerated. Feedings will be discontinued and an abdominal radiograph taken if there are any signs of feeding intolerance (recurrent emesis, gastric aspirate > 50% of previous feeding with abdominal distension or the presence of macroscopic blood in stools). In situations where feeds have been temporarily discontinued, patients may re-enter the study at the initiation of feeds. Patients who develop NEC may continue in the study if they are able to resume feeds after treatment. Inotropic support, if being weaned, is not a contraindication to begin or continue the protocol. Administration of probiotic will end at discharge, but the infant's status will continue to be monitored until 6 months post-discharge. Patient's participation in the study will end at 6 months post-discharge, or upon the death of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the NICU
* Written parental consent
* Birth weight < 2000 grams
* Hemodynamically stable
* < 48 hours of age

Exclusion Criteria:

* Evidence or suspicion of congenital intestinal obstruction or perforation
* Prenatal or postnatal diagnosis of gastroschisis, large omphalocele, or congenital diaphragmatic hernia
* Major congenital heart defects
* Anticipated transfer to a NICU not involved in the study

Ages: 1 Minute to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 751 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Number of deaths and episodes of nosocomial sepsis among probiotic exposed and non-exposed preterm infants | From birth to discharge from the NICU or death. Average time 2 months.
  Premature infants randomized within the first 48 hours of birth will be followed prospectively to determine number of deaths and episodes of nosocomial sepsis between placebo and control groups.

SECONDARY OUTCOMES:
Number of episodes of necrotizing enterocolitis experienced by each premature infant randomized to probiotic exposure or to placebo | From birth to discharge from the NICU or death. Average time: 2 months
  Premature infants randomized to placebo or treatment within the first 48 hours of birth will be followed prospectively to determine number of necrotizing enterocolitis episodes experienced using a modification of Bells criteria for Stage 2.

CONTACTS AND LOCATIONS:
Overall Officials: Mario A Rojas, MD, MPH, Principal Investigator — Vanderbilt University; Juan M Lozano, MD, Msc, Principal Investigator — Universidad Javeriana
Locations (8):
- Colombia (8):
  - Hospital San Vicente de Paul, Medellín, Antioquia
  - Hospital San Ignacio, Universidad Javeriana, Bogota, Cundinamarca
  - Policlinico del Olaya, Bogota, Cundinamarca
  - Clinica San Luis, Bucaramanga, Santander Department
  - Hospital Universitario de Santander, Bucaramanga, Santander Department
  - Clinica los Farallones, Cali, Valle del Cauca Department
  - Clinica Los Remedios, Cali, Valle del Cauca Department
  - Fundacion Valle de Lilli, Cali, Valle del Cauca Department

REFERENCES:
- [Derived] Rojas MA, Lozano JM, Rojas MX, Rodriguez VA, Rondon MA, Bastidas JA, Perez LA, Rojas C, Ovalle O, Garcia-Harker JE, Tamayo ME, Ruiz GC, Ballesteros A, Archila MM, Arevalo M. Prophylactic probiotics to prevent death and nosocomial infection in preterm infants. Pediatrics. 2012 Nov;130(5):e1113-20. doi: 10.1542/peds.2011-3584. Epub 2012 Oct 15. PMID 23071204